CLINICAL TRIAL: NCT04129606
Title: Bladder Perforation Post-TURBT: Definition, Incidence and Natural History. A Prospective Cohort Study
Brief Title: Bladder Perforation Post-TURBT: Definition, Incidence and Natural HistoryStudy
Acronym: TURBT-BP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abdelwahab Hashem (Other)
Responsible Party: Sponsor-Investigator, Abdelwahab Hashem, Principal Investigator, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TURBT-BP
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Bladder Cancer; Bladder Urothelial Carcinoma; Trauma; Injuries; Perforation of Bladder; Recurrence Tumor; Resection Margin; Seeding, Neoplasm
Keywords: Perforation of Bladder; Bladder Cancer; Resection Margin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Wounds and Injuries; Recurrence; Margins of Excision; Neoplasm Seeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TURBT (Other): Transurethral resection of bladder tumour
  Interventions: Diagnostic Test: Computed tomographic cystography

INTERVENTIONS:
Diagnostic Test: Computed tomographic cystography — CT cystogram performed after the procedure by the injection of 400mL of 1/4 saline-diluted contrast solution (meglumine ioxitalamate) with low-pressure infusion (60 cm gravity pressure) through the Foley catheter.
  Other Names: CT cystography

SUMMARY:
In view of sparse data of precise definition, risk factors, natural history and management of bladder perforation following Transurethral resection of bladder tumour (TURBT). We aim to correlate the relation between the site, depth and extent of resection with bladder perforation. Also, correlation between vertical depth, horizontal extent of resection and recurrence and progression of tumor

ELIGIBILITY:
Inclusion Criteria:

* papillary bladder tumor (denovo or recurrent)
* resectable nodular bladder tumor

Exclusion Criteria:

* Refuse to complete study requirements
* muscle invasive bladder tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of bladder perforation post-Transurethral resection of bladder tumour | 24 months
  calculate the numbers of bladder perforation diagnosed by CT cystogram divided by the total number of patients

SECONDARY OUTCOMES:
Correlation between the cystoscopical and radiological bladder perforation | 24 months
  compare the numbers of bladder perforation diagnosed by CT cystogram by the number of bladder perforation described by surgeon
assess the recurrence free rate in bladder perforation groups at 2 year follow up | 24 months
  calculate the number of recurrence pf bladder tumor in bladder perforation at 2 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Nasr Eltabey, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt